CLINICAL TRIAL: NCT01817062
Title: Retrospective Analysis of Intraoperative Volume Administration in Neonates Without Congenital Malformations With Very Low Birth Weight and Acute Abdomen.
Brief Title: Neonates With Very Low Birth Weight and Surgery Therapy of Acute Abdomen
Acronym: NeoNec
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, CVK and CCM, Charite University, Berlin, Germany
Other Study IDs: NeoNec
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Very Low Birth Weight
Keywords: Capillary leakage; Acute Abdomen; Low birth weight
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonates: Neonates with very low birth weight and surgery therapy of acute abdomen

SUMMARY:
Objective:

Due to high mortality rates the capillary leakage and the acute abdomen are important risk factors of the probability of survival. The aim of an optimal therapy of the acute abdomen within the neonatal period is beside the cure of the underlying disease the prophylaxis of capillary leakage with the help of optimised intra- and postoperative volume therapy.

Question:

Do the neonates with very low birth weight and a surgery therapy of acute abdomen benefit from early increase of the haemoglobin/haematocrit by optimised volume therapy with crystalloid and colloidal volume as prophylaxis of the capillary leakage?

ELIGIBILITY:
Inclusion criteria:

* All Children with very low birth weight who have undergone surgery of acute abdomen within the neonatal period between 2001 and 2011 on "Campus Charité Mitte" or "Charité Virchow - Klinikum".
* Neonates (calculated date of birth + 4 weeks)

Exclusion criteria:

* Birth weight > 1500g

Ages: 1 Minute to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with very low birth weight and surgery therapy of acute abdomen
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2001-01; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Capillary Leakage | 48 hours from Baseline (Operation)
  Postoperative Capillary Leakage (defined as weight gain within 48 hours or development of oedema within 48 hours)

SECONDARY OUTCOMES:
Amount of transfusions during surgery | Up to 5 hours
Re-surgery rate | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Length of stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Mortality | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - University Berlin, Berlin, State of Berlin, Germany